CLINICAL TRIAL: NCT07356284
Title: Emergent Large Vessel Occlusion Endovascular Rescue Therapy With Underlying Intracranial Stenosis
Acronym: EVEREST
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ProMedica Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EVEREST
Record Dates: First submitted 2026-01-20; First posted 2026-01-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Brain Stroke; Stenting Treatment; Acute Ischemic Stroke
Keywords: mechanical thrombectomy; Acute Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Randomized to Mechanical Thrombectomy (MT) plus adjunct Stenting (Experimental): Patients will have mechanical thrombectomy (MT) and stenting
  Interventions: Procedure: Mechanical Thrombectomy plus adjunct stenting
- Randomized to Mechanical Thrombectomy (MT) (Active Comparator): Patients will only have mechanical thrombectomy (MT) done
  Interventions: Device: Mechanical Thrombectomy

INTERVENTIONS:
Procedure: Mechanical Thrombectomy plus adjunct stenting — Mechanical thrombectomy and adjunct stentiing
  Other Names: mechanical thrombectomy; Stenting
  Arms: Randomized to Mechanical Thrombectomy (MT) plus adjunct Stenting
Device: Mechanical Thrombectomy — Mechanical thrombectomy only
  Arms: Randomized to Mechanical Thrombectomy (MT)

SUMMARY:
The study objective is to establish the safety and efficacy of endovascular adjunct stenting for patients undergoing mechanical thrombectomy (MT) that are found to have residual stenosis (70-99%) following attempted clot retrieval with either aspiration catheters or stent retrievers, per device instructions for use and device labeling.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age
2. Presenting with symptoms consistent with AIS
3. Imaging evidence of an anterior occlusion of the Internal Carotid Artery (ICA) or Middle Cerebral Artery Main Stem (MCA M1), or proximal M2 segment AND residual 70-99% stenosis of the index artery following attempted clot retrieval with either aspiration catheters or stent retrievers, per device instructions for use and device labeling
4. NIHSS ≥ 6
5. Ability to randomize within 24 hours of stroke onset.
6. Pre-stroke mRS score 0-2
7. Ability to obtain signed informed consent.
8. ASPECTS Score ≥ 6 by non-contrast CT scan
9. Score-ICAD score of ≥11 points at screening and/or persistent stenotic occlusion of ≥70% after MT
10. If indicated, thrombolytic therapy shall be initiated per the institution's usual care and the most recent version of the AHA/ASA Guidelines. Subjects eligible for IV thrombolysis should receive it without delay.
11. For subjects presenting >6 hours from stroke onset, infarct core volume <50 cc quantified by CTP

Exclusion Criteria:

1. Females who are pregnant, or those of child-bearing potential with positive urine or serum beta Human Chorionic Gonadotropin (HCG) test
2. Known severe allergy (more than a rash) to contrast media uncontrolled by medications.
3. CT evidence of the following conditions:

   * Midline shift or herniation
   * Evidence of intracranial hemorrhage
   * Mass effect with effacement of the ventricles
4. Acute bilateral strokes
5. Contraindication to antiplatelet (aspirin, clopidogrel, ticagrelor, cangrelor) or contrast agents
6. Intracranial tumors other than small meningioma, that do not require surgery for at least one year post randomization. Small meningioma is defined as a lesion measuring ≤20mm in maximum diameter or ≤4cm3 in volume, with no associated mass effect, peritumoral edema, or progressive neurological symptoms
7. Known hemorrhagic diathesis, coagulation factor deficiency, or on anticoagulant therapy with an International Normalized Ratio (INR) of >3.0 or Partial Thromboplastin Time (PTT) >3 times of normal
8. Baseline platelet count <80,000 per microliter (µl)
9. Life expectancy less than one year prior to stroke onset
10. Participation in another randomized clinical trial that could confound the evaluation of the study outcomes.
11. Any other condition (in the opinion of the site investigator) that precludes an endovascular procedure or poses a significant hazard to the patient if an endovascular procedure was performed
12. New diagnosis of atrial fibrillation or a history of atrial fibrillation
13. Suspected device-induced vasospasm defined as smooth transient narrowing of the target vessel
14. Vessel dissection including any of the following: presence of dissection flap, false lumen, contrast stagnation in the vessel wall, and/or improving stenosis

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 90 (+/- 30) days post treatment
  • Utility weighted 90-day Modified Rankin Score (mRS)
Primary Safety Endpoint | 90 (+/- 30 ) days post treatment
  Rate of symptomatic intracranial hemorrhage (sICH: Parenchymal hematoma Type 2 (PH2) with ≥4 points NIHSS worsening) at 24 hours (-12/+16 hours) from randomization)

SECONDARY OUTCOMES:
Secondary Safety Endpoint | 8 (+/- 3) days or Discharge post treatment
  Any neurological deterioration with ≥4 points worsening on NIHSS before discharge and unrelated to sICH or sedation (In addition to the routine 24-hour CT/Magnetic Resonance Imaging (MRI) scan, repeat neuroimaging is mandatory for any subsequent neurological deterioration at any time during hospitalization).
Secondary Safety Endpoint | Immediate post treatment
  Embolization into new territory (ENT)
Secondary Safety Endpoint | Immediate post treatment
  Distal embolization (DE)
Secondary Safety Endpoint | Immediate post treatment
  Major vessel injury (perforation, dissection)
Secondary Safety Endpoint | 1 year (+/- 60) days post treatment
  Ipsilateral recurrent stroke in the territory of the index artery from Day 1 through 1-year
Secondary Safety Endpoint | Immediate post treatment
  Rates of stent re-stenosis and stent thrombosis at the end of endovascular procedure
Secondary Safety Endpoint | 1 year (+/- 60) days post treatment
  • Intracranial stent stenosis (WASID) and stent thrombosis at any time between Day 1 to one year follow up
Secondary Safety Endpoint | 1 year (+/- 60) days post treatment
  Intracranial reintervention between Day 1 through 1-year (Any intervention or reintervention will be captured during that period)
Secondary Safety Endpoints | 1 year (+/- 60) days post treatment
  Neurological and All-Cause Mortality at 90 days and 1-year
Secondary Safety Endpoint | 1 year (+/- 60) days post treatment
  All serious adverse events (SAE), including serious adverse device events (SADE), serious adverse procedural events (SAPE), and unanticipated SAE.

OTHER OUTCOMES:
Secondary Efficacy Endpoints | 1 year (+/-60) days post treatment
  Utility weighted one-year Modified Rankin Score (mRS)
Secondary Efficacy Endpoints | 90 (+/-30) days post treatment
  90-day and one-year mRS ordinal shift (mRS 5 and 6 combined)
Secondary Efficacy Endpoints | 1 year (+/- 60) days post treatment
  90-day and one-year dichotomized mRS 0-2 outcome
Secondary Efficacy Endpoints | 1 year (+/-60) days post treatment
  90-day and one-year dichotomized mRS 0-3 outcome
Secondary Efficacy Endpoints | Immediate post treatment
  Change in NIHSS at 24 hours (12-40 hours hours) from randomization
Secondary Efficacy Endpoints | Day 8 (+/-3) days or discharge post treatment
  Change in NIHSS
Secondary Efficacy Endpoints | Day 8 (+/-) 3 days post treatment
  NIHSS of 0-2 or improvement of 8 or more points
Secondary Efficacy Endpoints | Immediately post treatment
  Rate of substantial reperfusion in the treatment arm at the end of procedure as TICI2b50 and TICI2b67 or higher
Secondary Efficacy Endpoints | Immediate post treatment
  Procedural/time metrics: Door to qualifying image, Image to Puncture, Puncture to mTICI 2b-3, Puncture to end of the procedure (defined as the final angiogram on the affected hemisphere)
Secondary Efficacy Endpoints | Day 8 (+/- 3) days post treatment
  Length of hospital stay
Secondary Efficacy Endpoints | 1 year (+/-60) days post treatment
  Effectiveness of stenting as measured by % stenosis within the MT adjunct stenting arm

CONTACTS AND LOCATIONS:
Overall Officials: Sami Al Kasab, MD, Principal Investigator — Medical University of South Carolina; Mouhammad Jumaa, MD, Principal Investigator — ProMedica Toledo Hospital; Tanya Siddiqui, Study Director — ProMedica Health System

IPD SHARING:
Plan to Share IPD: No